CLINICAL TRIAL: NCT03389906
Title: Inflammation Impact on Pain in Patients With Knee Osteoarthritis
Brief Title: Inflammation Impact on Pain in Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sten Rasmussen, MD, PhD (Other)
Collaborators: Aalborg University (Other)
Responsible Party: Sponsor-Investigator, Sten Rasmussen, MD, PhD, Professor Head of Department of Clinical Medicine, Northern Orthopaedic Division, Denmark
Organization: Northern Orthopaedic Division, Denmark (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: N-20160045
Record Dates: First submitted 2017-12-27; First posted 2018-01-04 (Actual); Last update posted 2021-08-12 (Actual); Status verified 2021-08

CONDITIONS: Inflammation; Osteo Arthritis Knee
MeSH Terms: conditions — Inflammation | interventions — Gold

STUDY DESIGN:
Intervention Model Description: Pilot study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Gold (Experimental): Approximately 72000, 20-40 my-meter diameter, sterilised gold particles (=20 mg) will be provided in vials (The Berlock® Gold Implants).
  Interventions: Other: Gold

INTERVENTIONS:
Other: Gold — Approximately 72000, 20-40 my-meter diameter, sterilised gold particles (=20 mg) will be provided in vials (The Berlock® Gold Implants). 5-10 ml of synovial fluid is aspirated (20G needle) from most affected OA-knee. The vial of gold particles are mixed with the synovial fluid, and the mix of gold and synovial fluid is injected intra-articularly into the patients knee.

SUMMARY:
The aim of this study is to use gold particles as a model compound to modulate specifically and selectively the function of macrophages and mast cells and investigate how this modulates pain and pain sensitization in the osteoarthritic knee assessed by mechanistic pain assessment technologies

DETAILED DESCRIPTION:
Osteoarthritis (OA) of the knee and hip is the most common musculoskeletal joint disease worldwide. Although a major symptom of OA is chronic joint pain, which has a significant effect on patients' quality of life, the pain mechanisms remain largely unknown.

Recently, clinical studies have suggested the existence of a neuropathic component in OA pain [5]. Accumulating evidence has been indicating that painful OA patients show peripheral and central sensitization [3,16]. Quantitative sensory testing (QST) is a relevant way to assess peripheral and central sensitization in joint pain [9]. The majority of studies have administered mechanical stimuli, and the most commonly used modality have been pressure. A recent review concluded that that people with OA have lower Pressure Pain Thresholds (PPT), facilitated temporal summation and impaired conditioned (CPM) compared with healthy controls [5]. Also, recent evidence have link QST profiles to the development of chronic pain [29,38], which emphasises the importance of studying the central nervous system.

Inflammation markers have been correlated with the pain intensity [35], and systemic inflammation can leads to sensitization of peripheral nociceptors [1]. Recently it was reported that higher preoperative levels of TNF-α, MMP-13 and IL-6 in synovial fluid may indicate a smaller improvement in pain 2 years after TKR [15].

Injectable solutions of gold-thio-compounds have been used to treat rheumatoid arthritis for nearly 100 years [13,21]. Several studies suggest that gold ions reduces pain, joint swelling, inflammation, and increase joint motility [24,31,33]. Gold salt therapy (auranofin; RidauraR) has been vetted by the FDA and approved (May 1985) and recommended by the American College of Rheumatology as a Disease Modifying Anti Rheumatic Drug - DMARD (https://www.rheumatology.org).

Gold salts, whether injected or given orally, have been shown to be effective [33,37] in reducing joint pain. Studies report patients going to total remission [28] and others report a 30% reduction in symptoms [20,27]. In addition, Clark et al., 1997 [8] concluded in a Cochrane meta-analysis that systemic treatment with gold was highly effective compared to placebo.

The use of gold salt given systemically have been criticized, since when gold compounds are made to circulate systemically via the circulatory system after oral or parenteral administration, the gold ions reach essentially all tissues and organs. In some patients, organs that are not involved in the arthritic disease, such as the kidneys, liver, and skin are adversely affected by gold. About 30% of patients develop such remote-organ "side effects" and discontinue gold treatment [20]. In addition, newer drugs have been developed with efficacy almost equal to gold ions in many patients, and less toxic.

To overcome the toxicity, a method that captures the efficacy of the gold ions but eliminates the remote side effects have been developed[10,23]. Briefly, the method isolates the gold ions within the affected joints by injecting solid gold metal directly into the diseased joint, whereby a very slow dissolution and local diffusion deliver the therapeutic gold ions to affected areas within the joint. In this therapy, 99.99% pure gold implants are injected into the body.

Individual single beads are implanted with a 15-16 gauge needle based on an X-ray picture in deeply anesthetized animals close to the capsule of the affected joint(s) (videos www.goldtreat.com). Over 3000 dogs, and more than 100 horses have had this treatment for osteoarthritis at 50+ veterinary clinics and hospitals throughout Europe. (www.goldtreat.com ). Success rates of 50 - 70% are quoted (www.goldtreat.com), and a double-blind, placebo controlled study on dogs showed improvement in over 80% of the dogs, which continues for 18 months [18] as the gold particles remain in the joint[26].

The systemic concentration of released gold ions is low but clinically effective and because the gold ions do not spread in the organism, but instead stay local, the technique is safe [12]. The trials to date indicate that only one local application is needed to obtain lifelong clinical effect [12].

To date it is still debated how much the inflammation per se contributes to pain in osteoarthritis. A variety of studies have investigates various aspects such as synovitis but still no clear associations to pain have been found[30]. Many studies have attempted to modulate the effect of the inflammatory mediators on the pain receptors by e.g. interacting with the arachidonic acid pathways[4]. As such compounds have both peripheral and central effects it is difficult to use such compounds a specific modulators of specific local inflammatory processes. No compounds have so far been used to modulate selectively the local organelles specifically involved in the inflammatory processes of joint pain.

Gold particles seems as the only known method to obtain such a local effect on one specific element involved in the inflammatory process - the macrophages and the mast cells.

If a foreign object gets embedded in the body, macrophages will attack the object and digest it.

If the foreign object has a diameter bigger than 20 microns the macrophage cannot engulf it. Instead the macrophages create a membrane on the surface of the foreign body and starts a chemical attack in order to dissolve it.

If the foreign body consist of gold the macrophages will cause release of gold ions from the foreign body.

Gold ions, taken up by the macrophages, causes them to malfunction[10,11,23]. As the macrophage is 'conductor' of the inflammatory process it causes a drastic restraint of the inflammation and finally bring it to a stop[22,25]. The released gold ions will be taken up by the macrophages themselves, but also diffuse out into the surrounding tissue where they are taken up by other cells as well e.g. mast cells and other connective tissue cells[7,32]. When the gold ions accumulate in the secretory granules of mast cells it blocks histamine release and thereby decrease the local oedema and additionally suppresses pain.

The amount of bio-released gold ions are related to the intensity of inflammation. Only few gold ions are released in immunological nonreactive tissue. This means that if a local inflammation that has been treated with gold implants, the increase in macrophages will cause an immediate inhibition of the inflammation.

The combined effect of gold ions on macrophages and mast cells is together believed to causes the significant reduction in pain following treatment with metallic gold particles. If this principle can be validated it may provide important information for development of new and better treatments for e.g. joint pain.

Recently, Seifert et al.[34] called for studies providing new insights into the mode of action of gold ions and suggest investigating the effects on key mechanisms involved in arthritis or other inflammatory conditions.

ELIGIBILITY:
Inclusion Criteria:

* Knee OA diagnosed based on the American College of Rheumatology criteria, KL (Kellgren-Lawrence) X-ray grade ≧ 2, pain for > 3months, maximal pain intensity VAS (visual analogue scale) ≧ 5 (0-10 scale) for the most painful knee during the last week. Knee joint effusion that can be aspirated

Exclusion Criteria:

* Pregnancy
* Drug addiction defined as the use of cannabis, opioids or other drugs
* Previous neurologic, musculoskeletal or mental illnesses
* Lack of ability to cooperate
* Current use of medications that may affect the trial e.g. analgesics, anti-inflammatory drugs
* Recent history of acute pain affecting the lower limb and/or trunk
* Past history of a chronic pain condition
* Participation in other pain trials throughout the study period

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2018-12-01 (Actual); Study Completion 2020-12-01 (Actual)

PRIMARY OUTCOMES:
WOMAC | 8 weeks, 2 years
  The WOMAC[6] is a subject-rated instrument that measures Osteoarthritis (OA)

SECONDARY OUTCOMES:
Quantitative sensory testing | 8 weeks
  Pressure Pain Sensitivity Cuff Pressure Algometry
Weekly pain diary | 8 weeks
  Subjects rated their pain intensity on a VAS scale every day at home. On the VAS scale ''0" indicates ''no pain", and ''10" indicates ''maximal pain".
  Subjects rated the pain severity for:
  Average Pain Score (APS) for the last 24 hours Worst pain for the last 24 hours Pain severity at night.
Inflammatory markers | 8 weeks
  Proteomic analysis of blood and synovial fluid
PainDetect questionnaire (PD-Q | 8 weeks, 2 years
  The PD-Q is a validated, easy to use screening tool that predicts the likelihood of a neuropathic pain component in chronic pain disorders[14]. It shows higher sensitivity and specificity in comparison with other neuropathic pain screening questionnaires. The questionnaire is comprised of 3 major components: gradation of pain, pain course pattern and radiating pain. There are 7 questions evaluating gradation of pain. Each question is scored by the patient using a 0 to 5 score with 0 = never, 1 = hardly notice, 2 = slightly, 3 = moderately, 4 = strongly and 5 = very strongly. There is one question evaluating pain course pattern. Patients select from one of four pictures to indicate which pattern of pain best describes their course of pain. Each picture is associated with a unique score of 0, -1, or +1 (2 pictures have this score possible). There is one question evaluating radiating pain with a yes (score of +2) or no (score of 0) response option.
Global Rating of Change Scale | 2 years
  we asked the question, "Concerning your knee, how will you describe yourself compared to immediately before injection of gold into your knee" and evaluated the answer at an 11-point scale from very much worse (-5) to complete recovered (5).

CONTACTS AND LOCATIONS:
Overall Officials: Lars Arendt-Nielsen, MD, PhD, Study Chair — Aalborg University
Locations (1):
- Aalborg University Hospital, Aalborg, Denmark

IPD SHARING:
Plan to Share IPD: Yes
Inflammatory markers may be shared with other researchers
Supporting Information: Study Protocol, SAP, ICF
Time Frame: After publication information is available.
Access Criteria: At the reasonable request to Sten Rasmusssen. (sten.rasmussen@rn.dk;s_rasmussen@dcm.aau.dk

REFERENCES:
- [Background] Turk DC, Dworkin RH, Allen RR, Bellamy N, Brandenburg N, Carr DB, Cleeland C, Dionne R, Farrar JT, Galer BS, Hewitt DJ, Jadad AR, Katz NP, Kramer LD, Manning DC, McCormick CG, McDermott MP, McGrath P, Quessy S, Rappaport BA, Robinson JP, Royal MA, Simon L, Stauffer JW, Stein W, Tollett J, Witter J. Core outcome domains for chronic pain clinical trials: IMMPACT recommendations. Pain. 2003 Dec;106(3):337-345. doi: 10.1016/j.pain.2003.08.001. PMID 14659516
- [Result] Andrew D, Greenspan JD. Mechanical and heat sensitization of cutaneous nociceptors after peripheral inflammation in the rat. J Neurophysiol. 1999 Nov;82(5):2649-56. doi: 10.1152/jn.1999.82.5.2649. PMID 10561434
- [Result] Arendt-Nielsen L, Egsgaard LL, Petersen KK, Eskehave TN, Graven-Nielsen T, Hoeck HC, Simonsen O. A mechanism-based pain sensitivity index to characterize knee osteoarthritis patients with different disease stages and pain levels. Eur J Pain. 2015 Nov;19(10):1406-17. doi: 10.1002/ejp.651. Epub 2014 Dec 29. PMID 25545011
- [Result] Arendt-Nielsen L, Nie H, Laursen MB, Laursen BS, Madeleine P, Simonsen OH, Graven-Nielsen T. Sensitization in patients with painful knee osteoarthritis. Pain. 2010 Jun;149(3):573-581. doi: 10.1016/j.pain.2010.04.003. Epub 2010 Apr 24. PMID 20418016
- [Result] Arendt-Nielsen L, Egsgaard LL, Petersen KK. Evidence for a central mode of action for etoricoxib (COX-2 inhibitor) in patients with painful knee osteoarthritis. Pain. 2016 Aug;157(8):1634-1644. doi: 10.1097/j.pain.0000000000000562. PMID 27007068
- [Result] Arendt-Nielsen L, Skou ST, Nielsen TA, Petersen KK. Altered Central Sensitization and Pain Modulation in the CNS in Chronic Joint Pain. Curr Osteoporos Rep. 2015 Aug;13(4):225-34. doi: 10.1007/s11914-015-0276-x. PMID 26026770
- [Result] Bellamy N, Buchanan WW, Goldsmith CH, Campbell J, Stitt LW. Validation study of WOMAC: a health status instrument for measuring clinically important patient relevant outcomes to antirheumatic drug therapy in patients with osteoarthritis of the hip or knee. J Rheumatol. 1988 Dec;15(12):1833-40. PMID 3068365
- [Result] Christensen MM, Danscher G, Ellermann-Eriksen S, Schionning JD, Rungby J. Autometallographic silver-enhancement of colloidal gold particles used to label phagocytic cells. Histochemistry. 1992;97(3):207-11. doi: 10.1007/BF00267629. PMID 1563970
- [Result] Clark P, Tugwell P, Bennet K, Bombardier C, Shea B, Wells G, Suarez-Almazor ME. Injectable gold for rheumatoid arthritis. Cochrane Database Syst Rev. 2000;1997(2):CD000520. doi: 10.1002/14651858.CD000520. PMID 10796386
- [Result] Courtney CA, Kavchak AE, Lowry CD, O'Hearn MA. Interpreting joint pain: quantitative sensory testing in musculoskeletal management. J Orthop Sports Phys Ther. 2010 Dec;40(12):818-25. doi: 10.2519/jospt.2010.3314. Epub 2010 Oct 22. PMID 20972347
- [Result] Danscher G. In vivo liberation of gold ions from gold implants. Autometallographic tracing of gold in cells adjacent to metallic gold. Histochem Cell Biol. 2002 May;117(5):447-52. doi: 10.1007/s00418-002-0400-8. Epub 2002 Apr 13. PMID 12029492
- [Result] Danscher G, Stoltenberg M. Silver enhancement of quantum dots resulting from (1) metabolism of toxic metals in animals and humans, (2) in vivo, in vitro and immersion created zinc-sulphur/zinc-selenium nanocrystals, (3) metal ions liberated from metal implants and particles. Prog Histochem Cytochem. 2006;41(2):57-139. doi: 10.1016/j.proghi.2006.06.001. Epub 2006 Aug 7. PMID 16949439
- [Result] Forestier J. Rheumatoid arthritis and its treatment by gold salts. The lancet 1934;224:646-648.
- [Result] Freynhagen R, Baron R, Gockel U, Tolle TR. painDETECT: a new screening questionnaire to identify neuropathic components in patients with back pain. Curr Med Res Opin. 2006 Oct;22(10):1911-20. doi: 10.1185/030079906X132488. PMID 17022849
- [Result] Gandhi R, Santone D, Takahashi M, Dessouki O, Mahomed NN. Inflammatory predictors of ongoing pain 2 years following knee replacement surgery. Knee. 2013 Oct;20(5):316-8. doi: 10.1016/j.knee.2012.10.015. Epub 2012 Nov 14. PMID 23157967
- [Result] Graven-Nielsen T, Wodehouse T, Langford RM, Arendt-Nielsen L, Kidd BL. Normalization of widespread hyperesthesia and facilitated spatial summation of deep-tissue pain in knee osteoarthritis patients after knee replacement. Arthritis Rheum. 2012 Sep;64(9):2907-16. doi: 10.1002/art.34466. PMID 22421811
- [Result] Guy W, Bonato RR. Manual for the ECDEU assessment battery. : US Department of Health, Education, and Welfare, National Institute of Mental Health, 1970
- [Result] Jaeger GT, Larsen S, Soli N, Moe L. Two years follow-up study of the pain-relieving effect of gold bead implantation in dogs with hip-joint arthritis. Acta Vet Scand. 2007 Mar 23;49(1):9. doi: 10.1186/1751-0147-49-9. PMID 17381835
- [Result] Jinks C, Jordan K, Croft P. Osteoarthritis as a public health problem: the impact of developing knee pain on physical function in adults living in the community: (KNEST 3). Rheumatology (Oxford). 2007 May;46(5):877-81. doi: 10.1093/rheumatology/kem013. Epub 2007 Feb 17. PMID 17308312
- [Result] Jones G, Brooks PM. Injectable gold compounds: an overview. Br J Rheumatol. 1996 Nov;35(11):1154-8. doi: 10.1093/rheumatology/35.11.1154. PMID 8948305
- [Result] Kean TA. Rheumatoid Arthritis and Gold Salts Therapy. Ulster Med J. 1934 Oct;3(4):284-9. No abstract available. PMID 20476023
- [Result] Labens R, Lascelles BD, Charlton AN, Ferrero NR, Van Wettere AJ, Xia XR, Blikslager AT. Ex vivo effect of gold nanoparticles on porcine synovial membrane. Tissue Barriers. 2013 Apr 1;1(2):e24314. doi: 10.4161/tisb.24314. PMID 24665389
- [Result] Larsen A, Kolind K, Pedersen DS, Doering P, Pedersen MO, Danscher G, Penkowa M, Stoltenberg M. Gold ions bio-released from metallic gold particles reduce inflammation and apoptosis and increase the regenerative responses in focal brain injury. Histochem Cell Biol. 2008 Oct;130(4):681-92. doi: 10.1007/s00418-008-0448-1. Epub 2008 Jun 10. PMID 18542984
- [Result] Lehman AJ, Esdaile JM, Klinkhoff AV, Grant E, Fitzgerald A, Canvin J; METGO Study Group. A 48-week, randomized, double-blind, double-observer, placebo-controlled multicenter trial of combination methotrexate and intramuscular gold therapy in rheumatoid arthritis: results of the METGO study. Arthritis Rheum. 2005 May;52(5):1360-70. doi: 10.1002/art.21018. PMID 15880810
- [Result] Leonaviciene L, Kirdaite G, Bradunaite R, Vaitkiene D, Vasiliauskas A, Zabulyte D, Ramanaviciene A, Ramanavicius A, Asmenavicius T, Mackiewicz Z. Effect of gold nanoparticles in the treatment of established collagen arthritis in rats. Medicina (Kaunas). 2012;48(2):91-101. Epub 2012 Apr 5. PMID 22491387
- [Result] Lie KI, Jaeger G, Nordstoga K, Moe L. Inflammatory response to therapeutic gold bead implantation in canine hip joint osteoarthritis. Vet Pathol. 2011 Nov;48(6):1118-24. doi: 10.1177/0300985810381910. Epub 2010 Sep 22. PMID 20861497
- [Result] Meier FM, Frerix M, Hermann W, Muller-Ladner U. Current immunotherapy in rheumatoid arthritis. Immunotherapy. 2013 Sep;5(9):955-74. doi: 10.2217/imt.13.94. PMID 23998731
- [Result] Menninger H, Herborn G, Sander O, Blechschmidt J, Rau R. A 36 month comparative trial of methotrexate and gold sodium thiomalate in the treatment of early active and erosive rheumatoid arthritis. Br J Rheumatol. 1998 Oct;37(10):1060-8. doi: 10.1093/rheumatology/37.10.1060. PMID 9825744
- [Result] Petersen KK, Arendt-Nielsen L, Simonsen O, Wilder-Smith O, Laursen MB. Presurgical assessment of temporal summation of pain predicts the development of chronic postoperative pain 12 months after total knee replacement. Pain. 2015 Jan;156(1):55-61. doi: 10.1016/j.pain.0000000000000022. PMID 25599301
- [Result] Petersen KK, Siebuhr AS, Graven-Nielsen T, Simonsen O, Boesen M, Gudbergsen H, Karsdal M, Bay-Jensen AC, Arendt-Nielsen L. Sensitization and Serological Biomarkers in Knee Osteoarthritis Patients With Different Degrees of Synovitis. Clin J Pain. 2016 Oct;32(10):841-8. doi: 10.1097/AJP.0000000000000334. PMID 26633689
- [Result] Rau R, Herborn G, Menninger H, Sangha O. Radiographic outcome after three years of patients with early erosive rheumatoid arthritis treated with intramuscular methotrexate or parenteral gold. Extension of a one-year double-blind study in 174 patients. Rheumatology (Oxford). 2002 Feb;41(2):196-204. doi: 10.1093/rheumatology/41.2.196. PMID 11886970
- [Result] Sadauskas E, Jacobsen NR, Danscher G, Stoltenberg M, Vogel U, Larsen A, Kreyling W, Wallin H. Biodistribution of gold nanoparticles in mouse lung following intratracheal instillation. Chem Cent J. 2009 Nov 20;3:16. doi: 10.1186/1752-153X-3-16. PMID 19930546
- [Result] Sanders M. A review of controlled clinical trials examining the effects of antimalarial compounds and gold compounds on radiographic progression in rheumatoid arthritis. J Rheumatol. 2000 Feb;27(2):523-9. PMID 10685827
- [Result] Seifert O, Matussek A, Sjogren F, Geffers R, Anderson CD. Gene expression profiling of macrophages: implications for an immunosuppressive effect of dissolucytotic gold ions. J Inflamm (Lond). 2012 Nov 9;9(1):43. doi: 10.1186/1476-9255-9-43. PMID 23140489
- [Result] Sturmer T, Brenner H, Koenig W, Gunther KP. Severity and extent of osteoarthritis and low grade systemic inflammation as assessed by high sensitivity C reactive protein. Ann Rheum Dis. 2004 Feb;63(2):200-5. doi: 10.1136/ard.2003.007674. PMID 14722211
- [Result] Williams HJ. Comparisons of sulfasalazine to gold and placebo in the treatment of rheumatoid arthritis. J Rheumatol Suppl. 1988 Sep;16:9-13. PMID 2903928
- [Result] Wylde V, Sayers A, Lenguerrand E, Gooberman-Hill R, Pyke M, Beswick AD, Dieppe P, Blom AW. Preoperative widespread pain sensitization and chronic pain after hip and knee replacement: a cohort analysis. Pain. 2015 Jan;156(1):47-54. doi: 10.1016/j.pain.0000000000000002. PMID 25599300
- [Derived] Rasmussen S, Petersen KK, Aboo C, Andersen JS, Skjoldemose E, Jorgensen NK, Stensballe A, Arendt-Nielsen L. Intra-articular injection of gold micro-particles with hyaluronic acid for painful knee osteoarthritis. BMC Musculoskelet Disord. 2024 Mar 12;25(1):211. doi: 10.1186/s12891-024-07321-4. PMID 38475764